CLINICAL TRIAL: NCT01957098
Title: The Effects of L-Arabinose and D-xylose on Intestinal Sucrase Activity in Man
Acronym: M192
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danisco (Industry)
Responsible Party: Principal Investigator, AAstrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: (KF) 11 324909
Record Dates: First submitted 2013-08-08; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Insulin Resistance
Keywords: L-arabinose; D-xylose; sucrose; glucose; insulin; C-peptide; GLP-1
MeSH Terms: conditions — Insulin Resistance | interventions — Pentoses; Xylose; Arabinose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0% pentose (Placebo Comparator): Pure sucrose without pentoses added.
  Interventions: Dietary Supplement: Placebo comparator: 0% pentose
- 4% D-xylose (Active Comparator): Sucrose drink supplemented with 4% D-xylose
  Interventions: Dietary Supplement: Active comparator: 4% D-xylose
- 8% D-xylose (Active Comparator): Sucrose drink supplemented with 8% D-xylose
  Interventions: Dietary Supplement: Active comparator: 8% D-xylose
- 8% L-arabinose (Active Comparator): Sucrose drink supplemented with 8% L-arabinose
  Interventions: Dietary Supplement: Active comparator: 8% L-arabinose

INTERVENTIONS:
Dietary Supplement: Placebo comparator: 0% pentose — 14 healthy subjects participated in a randomized double-blinded cross-over study based on four single tests. Sucrose containing drinks were supplemented with two different doses of D-xylose and in addition one dose of L-arabinose was included for comparison with earlier studies. Blood was collected fasting and for 3-h postprandially. Appetite sensations and energy intake were registered. Gastrointestinal symptoms were monitored for 24 hours
  Arms: 0% pentose
Dietary Supplement: Active comparator: 4% D-xylose
  Arms: 4% D-xylose
Dietary Supplement: Active comparator: 8% D-xylose
  Arms: 8% D-xylose
Dietary Supplement: Active comparator: 8% L-arabinose
  Arms: 8% L-arabinose

SUMMARY:
The purpose of this study is to investigate the effect of L-arabinose and D-xylose in a sugar-rich drink on intestinal sucrase activity in healthy volunteers by measuring postprandial blood glucose and insulin, and selected intestinal hormonal responses to increasing doses of L-arabinose and D-xylose.

DETAILED DESCRIPTION:
Based on previous scientific results we hypotesize, that pentoses decreases the demand for insulin in metabolizing a given dose of sucrose.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* BMI between 18.4-25 kg/m2
* age between 18 and 30

Exclusion Criteria:

* donation of blood 3 months before or during the study
* gastrointestinal disorders, diabetes, hypertension, hyperlipidemia, chronic infectious disease (HIV or hepatitis)
* smoking
* consumption of more than 21 alcoholic drinks/week
* elite athletes
* on medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose, insulin, C-peptide and GLP-1 | -15, 0, 15, 30, 45, 60, 90, 120, 180 min
  Level of glucose, insulin, C-peptide and glucagon-like peptide-1 (GLP-1) over time, the area under the curve (AUC), the peak value and time to peak

SECONDARY OUTCOMES:
Appetite measurements and energy intake | -15, 30, 60, 90, 120, 150 and 180 min
  Appetite measurements: area under/over the curve (AUC/AOC), 3-h mean. Energy intake: the ad libitum energy intake at lunch was registered. VAS was used to asses the palatability (appearance, smell, taste, after-taste and overall palatability) of the ad libitum lunch.

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Study Chair — University of Copenhagen
Locations (1):
- Institute of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark